CLINICAL TRIAL: NCT04423380
Title: A Phase I, Open-Label Study to Determine Safety, Tolerability, Pharmacokinetics (PK) and Preliminary Efficacy of SH3051 Capsule in Patients With Advanced Solid Tumors
Brief Title: A Study to Investigate Safety and Tolerability of SH3051 Capsule in Patients With Advanced Solid Tumors
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Nanjing Sanhome Pharmaceutical, Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SHC033-I-01
Record Dates: First submitted 2020-06-02; First posted 2020-06-09 (Actual); Last update posted 2020-06-09 (Actual); Status verified 2020-06

CONDITIONS: Advanced Solid Tumor
Keywords: advanced solid tumor; TGF-β RI; ALK5
MeSH Terms: interventions — Therapeutics

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- SH3051 capsules treatment (Experimental): Oral Twice Daily Administration of SH3051
  Interventions: Drug: SH3051 capsule treatment

INTERVENTIONS:
Drug: SH3051 capsule treatment — Starting dose 20mg,oral administered twice daily.If tolerated subsequent cohorts will test increasing doses (40mg,60mg,80mg,100mg) of SH3051.

SUMMARY:
The primary objective is to determine the safety profile of SH3051 in subjects with advanced solid tumors. The second objective is to evaluate the PK profile and preliminary efficacy of SH3051 solid tumors.

DETAILED DESCRIPTION:
This is a phase I, open-label study to assess the safety,tolerability, pharmacokinetics and preliminary efficacy of SH3051 capsule, a small molecule inhibitor of type I transforming growth factor-β(TGF-β) receptor serine/threonine kinase, in patients with advanced solid tumors.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 70 years inclusive;
* Histologically or cytologically confirmed advanced malignant solid tumors, eligible patients have failed standard treatment, have no standard treatment, or are not suitable for standard treatment at this stage as determined by the investigator.
* Must have at least one evaluable lesion in dose escalation period and one unidimensional measurable lesion according to RECIST version 1.1;
* Eastern Cooperative Oncology Group (ECOG) Performance Status of 0 or 1;
* Life expectancy ≥3 months;
* Adequate hematological and biological function, confirmed by the following laboratory values:ANC≥1.5×10^9/L;PLT≥75×10^9/L;Hb≥90g/L;TBIL≤1.5×ULN;AST and ALT≤3×ULN(ALT and AST≤5×ULN for subjects with liver cancer or hepatic metastases);CLcr>50 mL/min(according to Cockcroft-Gault);Child-Pugh score between 0~7 for subjects with primary hepatic carcinoma;APTT≤1.5×ULN;INR≤1.5×ULN.
* Men and women of childbearing potential are willing to employ an effective method of contraception for the entire duration of study and 6 months after the last dose, and female subjects of childbearing potential have a negative pregnancy test at baseline.
* Provision of signed and dated, written informed consent prior to any study-specific evaluation.

Exclusion Criteria:

* Previous treatment with any TGF-β inhibitors.
* Anticancer treatment including radiation therapy, chemotherapy, hormonal therapy, molecular targeted therapy, or immunotherapy within 4 weeks prior to the first dose of SH3051(use of mitomycin or nitrosoureas within 6 weeks prior to the first dose;use of oral oral fluorouracil and small molecule targeted drugs within 2 weeks ,or 5 half-lifes prior to the first dose;use of Chinese herbal anti-tumor treatment with 2 weeks prior to the first dose).
* Have systematic hormonal therapy(prednisone>20mg/d or similar drugs with equivalent dose)or immunosuppressor therapy with 14 days prior to the first dose of study drug, except using topical,ocular,intra-articular,intranasal,inhaled corticosteroids,and preventive therapy using corticosteroids in short period(for instance,to prevent hypersensitivity to contrast media).
* Participate in other clinical trials within 4 weeks prior to study entry.
* Concomitant use of any strong inhibitors or inducers of CYP3A4(except drug withdrawal within one week prior to first dose of study drug).
* History of allogeneic hematopoietic stem cell transplantation or organ transplantation.
* Adverse events occurred during previous anticancer therapy have not been recovered to ≤1(CTCAE 5.0)except toxicity with no significant risk determined by investigators such as alopecia.
* Evidence of central nervous system (CNS) metastases accompanied with clinical symptoms, or other evidence of uncontrolled CNS metastases Judged by investigators that the patient should not participate in the study.
* Presence of grade 3 or 4 gastrointestinal bleeding or esophageal and gastric varices.
* Have moderate or severe cardiac disease, including but not limited to severe arrhythmias or abnormal cardiac conduction, such as ventricular arrhythmias requiring clinical intervention, degree II-III atrioventricular block,QTcF≥450 ms for male, QTcF≥470 ms for female, or other structural heart disease with high risk as determined by investigators;history of acute coronary syndrome, congestive heart failure,aortic dissection,stroke or other≥grade 3 cardiovascular and cerebrovascular events within 6 months prior to the first dose of study drug;New York Heart Association (NYHA) Class II or greater heart failure, or LVEF<55%;cTnT or cTnI above the normal limit;NT-proBNP>1.25×ULN;uncontrolled hypertension;any risk factors to increase QTc or arrhythmias, including heart failure,hypokalemia,congenital long QTc syndrome,family history of long QT interval syndrome or history of unexplained sudden death occurred in first degree relative less than 40 years of age, or using any concomitant medication known to produce QTc prolongation.
* Have active infection requiring systemic with one week prior to the first dose the study drug.
* Infection with hepatitis B virus(HBV)and hepatitis C virus(HCV) (volunteers with HBsAg positive but HBV-DNA negative, or volunteers with HCV antibody positive but HCV-RNA negative can be enrolled).
* History of immune deficiency including HIV antibody positive.
* Major surgery(not include biopsy),or significant traumatism,or requiring selective operation within 4 weeks prior to study entry.
* Inability to swallow the drug, or severe gastrointestinal disease affecting absorption of the drug.
* Uncontrolled effusion in the third space, not suitable for entry as determined by the investigator.
* With alcohol or drug abuse disorder.
* With mental disorders or non-compliance.
* Women who are pregnancy or breastfeeding.
* Judgment by the investigator that the patient should not participate in the study.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2020-05-14 (Actual); Primary Completion 2021-03 (Estimated); Study Completion 2021-05 (Estimated)

PRIMARY OUTCOMES:
Maximum tolerated dose(MTD) | Within the first 28 days of consecutive treatment
Incidence of Dose Limiting Toxicity (DLT) | Within the first 28 days of consecutive treatment

SECONDARY OUTCOMES:
Area under the plasma concentration versus time curve(AUC)of SH3051 | 4 weeks
Elimination half-life(T1/2)of SH3051 | 4 weeks
Maximum(or peak)concentration of SH3051 | 4 weeks
Overall Response Rate(ORR) | up to 12 months
Progression-free survival(PFS) | up to 12 months
Disease control rates(DCR） | up to 12 months
Duration of response(DOR) | up to 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Jin Li, MD, Principal Investigator — Shanghai East Hospital
Locations (1):
- Shanghai East Hospital, Shanghai, China